CLINICAL TRIAL: NCT01342263
Title: Utilization of an Interactive Internet-based Platform for Managing Chronic Diseases at a Distance
Brief Title: Trial of an Internet-based Platform for Managing Chronic Diseases at a Distance
Acronym: iCDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Fraser University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Michael Smith Foundation for Health Research (Other)
Responsible Party: Principal Investigator, Scott Lear, Professor, Simon Fraser University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 711174
Record Dates: First submitted 2011-04-21; First posted 2011-04-27 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Ischemic Heart Disease; Heart Failure; Chronic Kidney Disease; Diabetes; Chronic Obstructive Pulmonary Disease
Keywords: Chronic disease management; Ischemic heart disease; Heart failure; Chronic kidney disease; Diabetes; Chronic obstructive pulmonary disease; Telehealth; Internet
MeSH Terms: conditions — Myocardial Ischemia; Heart Failure; Renal Insufficiency, Chronic; Diabetes Mellitus; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Does not get to participate in the interactive chronic disease website.
- iCDM (Experimental): The iCDM will support patient self-management through collaborative planning and goal setting, education and skill development, support for behaviour change, and regular patient monitoring with follow-up. For each chronic condition, we have outlined sample patient signs and symptoms to be monitored, frequency of patient provider contact and frequency of patient prompt questions on their condition. The main premise of the iCDM is that only those patients who generate 'alerts' will be contacted by the iCDM nurse allowing for the potential to manage more patients than through traditional means of required patient follow-up regardless of patient condition . Across these five diseases are the following cross-cutting features: nutrition therapy, exercise therapy, psychological support, medication adherence and smoking cessation.
  Interventions: Behavioral: iCDM

INTERVENTIONS:
Behavioral: iCDM — The iCDM intervention will be managed by a nurse with experience in chronic disease management who will review patient data, communicate with the patients, implement the Treatment Algorithms and interact with the patients' PCP. Patients will also be able to interact with a dietitian and exercise specialist to support them in their disease management. These personnel will have formal training in principles of the Transtheoretical Model of Change and Social Cognitive Theory.
  Arms: iCDM

SUMMARY:
In 2005, more then one-third of Canadians were burdened with one or more chronic diseases. Patients with one chronic disease often have, or are at risk for, another chronic disease. This group of complex patients represents a substantial challenge to healthcare resources. For patients in rural communities, the opportunity to attend ambulatory care clinics is not always an option. Additionally, the opportunity for rural patients to receive quality care close to, or within their homes, is of great benefit as it reduces the need for extensive travel and the potential burden of clinical visits. The use of telehealth has been identified as an effective modality for chronic disease management and is actively promoted by national organizations as having great promise for health service delivery in rural areas. The Internet as a mode for healthcare delivery has numerous advantages: 1. it is ubiquitous with increasing access in all age groups, 2. it is inexpensive, 3. it facilitates both patient data transfer and patient feedback, thereby supporting patient self-management, 4. it is scalable to large patient volumes, 5. it delivers health care directly to the patient and 6. it requires minimal set-up for patients with current Internet access.

The investigators propose to develop and evaluate a multi-chronic disease management program delivered through the Internet (with telephone supports) focused on high-impact chronic diseases targeted to patients in rural communities.

This study will consist of a single-blinded randomized controlled trial to investigate the efficacy of the iCDM in 318 patients with two or more of the target chronic diseases living in rural areas. Within this Aim, the investigators will be able to address the following research questions:

Q1. What is the effect of iCDM on healthcare utilization and patient self-management outcomes? Q2. What is the long-term compliance to the iCDM? Q3. What is the level of patient and provider satisfaction?

DETAILED DESCRIPTION:
A study population of men and women over 19 years will be identified through nurse practitioners, primary care networks, and other practicing primary care physicians located within the Northern Health, Fraser Health, Interior Health, Vancouver Island Health and Vancouver Coastal Health Authorities. Patients will be eligible if they have two or more of the five targeted chronic diseases; daily Internet access (home, work or other environment) by and means; and able to read, write and understand English without difficulty. A total of 318 patients (159 per group) will be recruited and randomized to either usual care, or a 24-month interactive chronic disease management program delivered via the Internet.

Usual Care Group Patients randomized to usual care will be given educational information regarding general chronic disease management and a list of Internet-based resources, and will return to the care of their primary care physician. Patients will be contacted after 24 months for an outcome assessment. There will be no contact between the study personnel and usual care patients for the duration of the study, nor will there be any attempt to control the level of patient care.

iCDM Experimental Group The iCDM is a 24-month interactive website that has been designed for patients with two or more of the following chronic diseases: ischemic heart disease, heart failure, diabetes, chronic kidney disease and chronic obstructive pulmonary disease. The iCDM is managed by a nurse with experience in chronic disease management who will review patient data, communicate with patients, implement treatment and interact with the patients' primary care physician. Patients will also be able to interact with a dietician and exercise specialist to support their disease management.

The main premise of the iCDM is that users will log-on on a regular basis and enter data related to how they are feeling and some physical measures (such as body weight, blood sugar, blood pressure, as relevant). Based on answers to these questions, the website may show a message either saying everything is fine or give a warning, informing the patient of their answers and that a nurse will be contacting them on the next business day. If the nurse receives an alert in his/her email inbox, he/she will telephone the patient within approximately 24 hours to discuss the entered data. The nurse may also direct the patient to discuss with the dietician or exercise specialist, or tell them that it is probably best for them to visit their physician for their symptoms.

Patients will have access to the iCDM for a 24 month period. Their family physician will receive a letter indicating their participation in the program and the conditions under which they may be contacted. At 24 months patients will be contacted for an outcome assessment.

ELIGIBILITY:
Inclusion Criteria:

* two or more of the following chronic diseases; heart disease, heart failure, chronic kidney disease, diabetes and COPD
* daily Internet access
* able to read, write and understand English

Exclusion Criteria:

* patients with significant co-morbidities that may interfere with effective management
* patients who have scheduled surgical procedures
* patients who are unable to provide informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2011-05; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Healthcare utilization | 24 months
  Hospital admissions, length of hospital stay, emergency room visits, physician visits, diagnostic and lab procedures.

SECONDARY OUTCOMES:
health-related Quality of life | 24 months
  Assessed by the Medical Outcomes Study 36-item Short Form survey.
Self-management | 24 months
  Assessed by the Health Education Impact Questionnaire (heiQ).
Social support | 24 months
  Assessed using the Medical Outcomes Study Social Support Scale.
Patient and Provider Experience and Satisfaction | 24 months
  Patients enrolled in the iCDM intervention and their family physicians will undergo a semi-structured, open-ended interview at the end of the intervention to explore patient experiences and to increase our understanding of patient factors that influence acceptance and use.
Adherence to the iCDM | 24 months
  Assessed through website use (logins) and completion of data entry.
Health outcomes | 24 months
  Assessed by the EuroQol EQ-5D-5L health questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Lear, PhD, Principal Investigator — Simon Fraser University
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Lear SA, Norena M, Banner D, Whitehurst DGT, Gill S, Burns J, Kandola DK, Johnston S, Horvat D, Vincent K, Levin A, Kaan A, Van Spall HGC, Singer J. Assessment of an Interactive Digital Health-Based Self-management Program to Reduce Hospitalizations Among Patients With Multiple Chronic Diseases: A Randomized Clinical Trial. JAMA Netw Open. 2021 Dec 1;4(12):e2140591. doi: 10.1001/jamanetworkopen.2021.40591. PMID 34962560